CLINICAL TRIAL: NCT06207500
Title: Impact of Routine Pharmacist-led Medication Reconciliation on Medication Discrepancies and Post-hospital Healthcare Utilisation
Brief Title: Evaluation of Pharmacist-led Medication Reconciliation Service Benefits in Hospitalised Medical Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID 19 declaration in Slovenia for the second time and subsequent reorganization of intervention ward
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Jošt, Clinical Pharmacist, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 8019163
Record Dates: First submitted 2023-12-22; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Medication Reconciliation
Keywords: medication error; unplanned healthcare utilisation; transitions of care; pharmacist; patient discharge; patient counselling

STUDY DESIGN:
Intervention Model Description: Pragmatic prospective controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Patients were offered pharmacist- led medication reconciliation on admission and discharge coupled with patient counselling.
  Interventions: Procedure: Pharmacist-led Medication Reconciliation
- Control Group (No Intervention): Patients received standard care - only written instructions on discharge medications in the discharge letter, according to the standard practice.

INTERVENTIONS:
Procedure: Pharmacist-led Medication Reconciliation — The best possible medication history (BPMH) at hospital admission was obtained from medical and pharmacy records and by interviewing the patient or carers. The BPMH - an accurate and complete (or as close as possible) list of medications the patient is currently taking - was documented in the medication information system. At hospital admission the BPMH was compared with the therapy in hospital to identify discrepancies. All discrepancies were discussed with the treating physician, unintentional discrepancies were reconciled. Intentional discrepancies were documented in the medical records. Prior to discharge from hospital, the BPMH and the medications planned in the discharge therapy were compared again to ensure that all unintentional discrepancies were corrected. Intentional discrepancies were explained in the discharge letter. Individual patient counselling on discharge medications and pharmacotherapy changes was conducted and coupled with written instructions in lay language.
  Arms: Intervention Group

SUMMARY:
Background:

Transitions of care often lead to medication errors and unnecessary healthcare utilisation. It has been repeatedly shown that medication reconciliation can at least partially reduce this risk.

Objective:

The aim of this prospective pragmatic trial was to evaluate the effectiveness of pharmacist-led medication reconciliation offered to medical patients as part of routine clinical practise.

The main questions to be answered were:

* the effectiveness of pharmacist-led medication reconciliation on medication discrepancies at discharge and 30 days after discharge
* the effectiveness of pharmacist-led medication reconciliation on healthcare utilisation within 30 days after discharge.

Participants in the intervention group were offered the following:

* medication reconciliation on admission
* medication reconciliation on discharge, coupled with patient counselling, provided by clinical pharmacists.

Participants in the control group were offered standard care.

DETAILED DESCRIPTION:
Design: pragmatic, prospective, controlled clinical trial

Setting: Five general medical wards at the University Clinic of Respiratory and Allergic Diseases in Slovenia:

* one intervention ward with a routine pharmacist-led medication reconciliation service
* four control wards

Data collection:

* Data collection and outcome assessment were performed by research pharmacists who were clinical pharmacists or final year clinical pharmacy residents not involved in the treatment of the included patients.
* Data for the assessment of medication errors at discharge were obtained from the patients' medical records and the study documentation.
* The reason for the patient's hospitalisation was obtained from the discharge letter and divided into acute or planned admissions. The main diagnosis was the reason for admission, while all other patient diagnoses listed were used to assess comorbidity.
* Patient comorbidity was assessed using the Charlson Comorbidity Index
* For patients in the control group the BPMH was collected in the same way as in the intervention group. However, it was only used for study purposes and was not documented in the patients' medical records
* Data on healthcare utilisation and medication discrepancies after hospital discharge were collected through patients or caregivers' phone interview.

ELIGIBILITY:
Inclusion Criteria:

* All adult medical patients admitted to the study wards

Exclusion Criteria:

* patients who do not speak Slovenian,
* transferred from another ward,
* previously included in the same study.

Subsequent exclusion from the analysis:

* patients hospitalised only for diagnostic purposes,
* patients transferred to another ward or hospital,
* patients that died during hospitalisation,
* patients from the control group who were offered medication reconciliation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Unplanned healthcare utilisation within 30 days after discharge | within 30 (±5) days after hospital discharge
  Unplanned healthcare utilisation within 30 days of hospital discharge was defined as any unplanned visit to a general practitioner, specialist, emergency department (ED), or hospitalisation or death. The visits were classified as unplanned, if sudden health problems required medical attention, and planned, if scheduled. Data on mortality due to any reason were also collected 30 days after discharge. For each patient, only the most detrimental outcome was classified.

SECONDARY OUTCOMES:
Serious unplanned healthcare utilisation within 30 days after discharge | within 30 (±5) days after hospital discharge
  Serious unplanned healthcare utilisation were defined as any unplanned ED visit or hospitalisation or death within 30 days from hospital discharge.
Clinically important medication errors at discharge | On the day of hospital discharge (up to 365 days from hospital admission)
  Unintentional discrepancies and undocumented intentional discrepancies between the therapy the patient was taking before admission (BMPH) and the therapy recommended in the discharge letter were defined as medication errors. Their clinical importance was assessed using a 4-point Likert scale ranging from not important, not very important, very important to life-threatening medication errors. Very important and life-threatening medication errors represent clinically important medication errors.
Medication discrepancies at 30 days | At 30 (±5) days after hospital discharge
  Medication discrepancies 30 (±5) days after hospital discharge were defined as the discrepancies between the discharge therapy and the therapy the patient was taking 30 (±5) days after hospital discharge.
  The discrepancies were defined as intentional if the patient intentionally took the therapy differently than recommended in the discharge letter. The reason for the discrepancy was also recorded - the patient's own informed decision or due to instructions from the treating physician (general practitioner, specialist).
  Unintentional discrepancies were defined as discrepancies from the therapy recommended in the discharge letter of which the patients were unaware. The clinical importance of unintentional discrepancies was assessed using a 4-point Likert scale, ranging from not important, not very important, very important, to life- threatening.
All healthcare utilisation within 30 days after discharge | within 30 (±5) days after hospital discharge
  Healthcare visits within 30 days of hospital discharge were defined as any visit to a general practitioner, specialist, emergency department (ED), or hospitalisation. These visits were classified as unplanned, if sudden health problems required medical attention, and planned, if scheduled. Data on mortality due to any reason were also collected 30 days after discharge. For each patient, only the most detrimental outcome was classified.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Respiratory and Allergic Diseases Golnik, Golnik, Select State, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jost M, Kerec Kos M, Kos M, Knez L. Effectiveness of pharmacist-led medication reconciliation on medication errors at hospital discharge and healthcare utilization in the next 30 days: a pragmatic clinical trial. Front Pharmacol. 2024 Mar 28;15:1377781. doi: 10.3389/fphar.2024.1377781. eCollection 2024. PMID 38606174